CLINICAL TRIAL: NCT03802721
Title: Pharmacokinetics of Benzo[a]Pyrene: Impact of Diet
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Lawrence Livermore National Laboratory (Other); Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Williams, Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LPI-8789; R01ES028600 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Environmental Exposure
Keywords: Benzo[a]pyrene; Accelerator Mass Spectrometry; Polycyclic Aromatic Hydrocarbons; cruciferous vegetable; Brussels sprouts; 3,3'-diindolylmethane; DIM; indole-3-carbinol; I3C; PAH

STUDY DESIGN:
Masking Description: Deidentified samples will be analyzed by AMS at Lawrence Livermore National Laboratory and the pharmacokinetics determine at Pacific Northwest National Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 50 ng dose; Brussels sprouts before 50 ng dose; DIM supplement before 50 ng dose (Experimental): Cycle 1: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Subjects will consume 50 g (about 1/2 cup) of lightly steamed Brussels sprouts each evening for 7 days prior to taking capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 3: Subjects will consume 300 mg DIM supplement ( 2 capsules of BioResponse DIM® 150) each evening for 7 days prior to taking capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP). A 300 mg DIM dose will be co-administrated with the 50 ng BaP dose.
  At least 3 weeks will pass between cycles as a washout period.
  Interventions: Drug: [14C]-benzo[a]pyrene; Drug: Brussels sprouts before 50 ng dose; Drug: DIM supplement before 50 ng dose

INTERVENTIONS:
Drug: [14C]-benzo[a]pyrene — Oral micro-dose (50 ng) (5.4 nCi)
  Other Names: Carcinogenic PAH environmental pollutant
Drug: Brussels sprouts before 50 ng dose — Brussels sprouts for 7 days before 50 ng (5.4 nCi) dose of BaP
  Other Names: Brussels sprouts and carcinogenic PAH
Drug: DIM supplement before 50 ng dose — DIM supplement for 7 days before 50 ng (5.4 nCi) dose of BaP and coadministration with DIM supplement
  Other Names: Cruciferous vegetable supplement and carcinogenic PAH

SUMMARY:
Evaluation of the pharmacokinetics for [14C]-benzo[a]pyrene ([14C]-BaP) and metabolites in plasma and urine over 48 hours following a 50 ng dose (5.4 nCi) alone, following 7 days' consumption of Brussels sprouts, and following 7 days' consumption of a supplement containing 3,3'-diindolylmethane (DIM).

DETAILED DESCRIPTION:
The pharmacokinetics for [14C]-BaP and metabolites will be assessed by UHLPC-Accelerator Mass Spectrometry (AMS, Lawrence Livermore National Laboratory) in plasma and urine collected over 48 hours following oral doses of 50 ng dose (5.4 nCi) alone, following 7 days' consumption of Brussels sprouts, and following 7 days' consumption of a supplement containing 3,3'-diindolylmethane (DIM).

The investigators hypothesize that pre-administration of Brussels sprouts or DIM will alter [14C]-BaP metabolism and increase the rate of elimination consistent with predictions based on a previously developed Physiologically-Based Pharmacokinetic (PBPK) model for BaP. Briefly, this hypothesis will be tested by dosing individuals with 50 ng [14C]-BaP alone and, following a 3-week washout period, ingestion of about 50 g Brussels sprouts or 300 mg of 3,3'-diindolylmethane (DIM) supplement for 7 days prior to the [14C]-BaP micro-dose. The impact of the supplement and the whole food will be assessed with respect to alterations in uptake from the GI tract, metabolism and rate of elimination. The consumption of cruciferous vegetables will be assessed at the beginning of the study by completion of a dietary questionnaire to examine typical eating patterns in the previous 3 months and by collection and extraction of blood and urine to assay for DIM by LC/ESI-MS/MS-SRM). In addition, for each phase, urine will be assayed for DIM as an estimate of crucifer or DIM supplement intake.

In preclinical and clinical studies, administration of Brussels sprouts or DIM impacts the activity of the same enzymes responsible for the phase 1 (CYP1A1 and CYP1B1) and phase 2 enzymes (GSTM1, UGT, SULT). Monitoring changes in β-estradiol metabolites will confirm the mechanism of alteration in the metabolic profile of [14C]-BaP.

Metabolite profiles and kinetics of elimination are predicted to be consistent with a BaP physiologically based pharmacokinetic (PBPK) model developed by Pacific Northwest National Laboratory (PNNL). A non-smoker, not exposed occupationally, receives 270-700 ng of BaP daily; about 95% dietary. The WHO has set an estimated safe daily lifetime (70 year/70 Kg individual, cancer endpoint) exposure to BaP of 42-350 ng. This protocol represents de minimus risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 (inclusive)
* If female, must be post-menopausal or have had surgical sterilization to eliminate any possibility for fetal exposure
* Willing to defer blood donation for one month before, throughout, and one month after completion of study activities
* Willing to avoid consuming cruciferous vegetables, I3C or DIM supplements, smoked or cured meat or cheeses, or charcoal-grilled meats for 2 weeks prior to and during each study cycle (gas grilled foods acceptable)
* Health history review and physical assessment showing general good health, as determined by study physician. Acceptable physical exam may have been conducted as part of protocol 8233 or 8554 if subject has not had significant changes in health status.

Exclusion Criteria:

* Smoker (tobacco or other substances) or use of smokeless tobacco in past 3 months or living with smoker
* Regular use of medications that affect gut motility or nutrient absorption (e.g. cholestyramine, sucralfate, orlistat, pro- or anti-motility agents)
* History of gastrointestinal surgery (e.g. bariatric surgery, cholecystectomy) or gastrointestinal disorder (Crohn's disease, celiac disease, IBS, or colitis)
* Current or history of kidney or liver disease
* Prior high-dose 14C exposure from medical tests. (micro-dose 14C exposure not exclusionary)
* Occupational PAH exposure (e.g. roofers, asphalt pavers, fire-fighters, etc.)
* Regular use of indole-3-carbinol or DIM dietary supplements
* Allergy or intolerance to Brussels sprouts or similar foods

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified samples sent to Lawrence Livermore National Laboratory Deidentified data sent to Pacific Northwest National Laboratory

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose: Cycle 1: Capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Subjects will consume 50 g (about 1/2 cup) of lightly steamed Brussels sprouts each evening for 7 days prior to taking capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 3: Subjects will consume 300 mg DIM supplement ( 2 capsules of BioResponse DIM® 150) each evening for 7 days prior to taking capsule containing 50 ng (5.4 nCi) [14C]-benzo[a]pyrene (BaP). A 300 mg DIM dose will be co-administrated with the 50 ng BaP dose.
  At least 3 weeks will pass between cycles as a washout period.
  [14C]-benzo[a]pyrene: Oral micro-dose (50 ng) (5.4 nCi)
  Brussels sprouts before 50 ng dose: Brussels sprouts for 7 days before 50 ng (5.4 nCi) dose of BaP
  DIM supplement before 50 ng dose: DIM supplement for 7 days before 50 ng (5.4 nCi) dose of BaP and coadministration with DIM supplement
Period: Overall Study
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of 14C-BaP Cmax
Description: Determination of highest concentration of 14C-BaP in plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine Cmax.
Time Frame: 0-48 hours for each of 3 dosing cycles, with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Number analyzed (Participants) | 7
fg [14C]-BaP/mL plasma
  50 ng [14C] BaP | 3.69 (4.12)
  Brussels sprouts before 50 ng [14C] BaP | 1.67 (1.03)
  DIM supplement before 50 ng [14C] BaP | 0.68 (0.51)

2. Secondary Outcome: Time at Highest Plasma Concentration of 14C-BaP Tmax
Description: Determination of time at which plasma concentration of 14C-BaP is highest. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine Tmax.
Time Frame: 0-48 hours for each of 3 dosing cycles, with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Number analyzed (Participants) | 7
hour
  50 ng [14C] BaP | 1.58 (1.16)
  Brussels sprouts before 50 ng [14C] BaP | 1.14 (0.90)
  DIM supplement before | 14.00 (19.17)

3. Secondary Outcome: Area Under Plasma Concentration of 14C-BaP Versus Time Curve AUC
Description: Integration of concentration of 14C-BaP in plasma over time. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine AUC.
Time Frame: 0-48 hours for each of 3 dosing cycles, with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma x hour
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Number analyzed (Participants) | 7
fg [14C]-BaP/mL plasma x hour
  50 ng [14C] BaP | 10.93 (9.19)
  Brussels sprouts before 50 ng [14C] BaP | 9.34 (10.02)
  DIM supplement before 50 ng [14C] BaP | 5.51 (6.17)

4. Secondary Outcome: Rate of Elimination of 14C-BaP (Half Life)
Description: Determination of constants for rate of elimination of 14C-BaP from plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine half-life.
Time Frame: 0-48 hours for each of 3 dosing cycles, with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
Number analyzed (Participants) | 7
hour
  50 ng [14C] BaP | 3.69 (3.80)
  Brussels sprouts before 50 ng [14C] BaP | 3.86 (4.62)
  DIM supplement before 50 ng [14C] BaP | 9.75 (13.25)

ADVERSE EVENTS:
Time Frame: 9 days for Brussels sprouts (BS) and DIM cycles- Participants were assessed for adverse events beginning beginning 7 days prior to the [14c]-BaP dose administration (time= 0 hour), when participants began consuming BS or DIM supplements. They were assessed until 0.25h after the final blood sample collection time point (time = 48 hour) and removal of the peripheral IV catheter. 48.5 h for BaP-only cycle - 0.25h prior to dose until 0.25 hr after final blood sample at 48 h.
Description: The definitions of adverse event and serious adverse event used to determine incidence are consistent with clinicaltrials.gov definitions. Each participant was verbally asked about the occurrence of adverse events at each clinical visit by the research nurse.
Arm/Group | 50 ng Dose; Brussels Sprouts Before 50 ng Dose; DIM Supplement Before 50 ng Dose
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03802721/Prot_SAP_ICF_000.pdf